CLINICAL TRIAL: NCT02486146
Title: GI Biorepository of Tissue and Bodily Fluids
Status: Completed | Type: Observational
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Other Study IDs: 575191
Record Dates: First submitted 2015-06-19; First posted 2015-07-01 (Estimated); Last update posted 2017-06-21 (Actual); Status verified 2017-06

CONDITIONS: Gastrointestinal Diseases
MeSH Terms: conditions — Gastrointestinal Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to establish the working protocols for a general biorepository with the specific aim of procuring tissues and bodily fluids from the human gastrointestinal tract from a diverse range of clinical patients at the UC Davis Medical Center. The establishment of a GI-specific biorepository will support future translational endeavors within the UC Davis campus by providing laboratories with readily available GI tissue and bodily fluid samples to test newly developed hypotheses with relative ease.

DETAILED DESCRIPTION:
UC Davis is currently lacking a general use biorepository for GI tissues and bodily fluids. As with any translational research study, the procurement of human tissue samples can be a difficult and time- consuming process. The establishment of this biorepository will help streamline GI biospecimen collection and centralize these samples in a conveniently located space to facilitate the implementation of future unspecified translational studies.

ELIGIBILITY:
Inclusion Criteria:

* all consenting adults aged 18 years or older with an appointment with a healthcare professional in the Division of Gastroenterology or the Department of Surgery

Exclusion Criteria:

* minors, pregnant women, prisoners, and all other vulnerable populations who are unable to consent.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals to be included will be all consenting adults aged 18 years or older with an appointment with a healthcare professional in the Division of Gastroenterology or the Department of Surgery. During their routinely scheduled appointment or procedure, eligible individuals will be informed of the program by the attending physician and encouraged to participate in order to establish a diverse collection of samples of GI-related pathologies and matched controls. The investigators' exclusion criteria will include minors, pregnant women, prisoners, and all other vulnerable populations who are unable to consent.
Sampling Method: Non-Probability Sample
Enrollment: 789 (Actual)
Dates: Start 2014-10; Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
To build a model biorepository to streamline the biobanking process and provide centralized specimens and associated health information for translational research. | 4 years
  To have biospecimens available for the UC Davis IRB approved studies.

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Jui Yvonne Wan, PhD, Principal Investigator — University of California, Davis
Locations (1):
- UC Davis Health System, Sacramento, California, United States